CLINICAL TRIAL: NCT02713464
Title: Effect of Education on Prevalence of Kernicterus in Five Regions in Nigeria
Brief Title: Does Maternal Instruction Prevent Kernicterus in Nigeria?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilimetrix s.r.l. (Other)
Collaborators: Jos University Teaching Hospital (Other); Bayern University Teaching Hospital (Unknown); Ahmadu Bello University Teaching Hospital (Other); Massey Street Children's Hospital (Other); Federal Medical Center Asaba (Unknown); University of Minnesota (Other)
Responsible Party: Principal Investigator, Richard Patridge Wennberg, Principal Investigator, Bilimetrix s.r.l.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SKIN1
Record Dates: First submitted 2016-03-12; First posted 2016-03-18 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Kernicterus
MeSH Terms: conditions — Kernicterus | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- maternal education (Active Comparator): Phase IIa: Pregnant women attending antenatal clinics or postpartum in clinics or hospital who receive programmed maternal education about risks and care of newborn jaundice.
  Interventions: Behavioral: maternal education
- Historic control (No Intervention): Phase I: (before-after design) Baseline prevalence of acute bilirubin encephalopathy before maternal education instituted.
- No intervention (No Intervention): Phase IIb: Opportunistic controls - infants of mothers who failed to receive education about risks and care of newborn jaundice.

INTERVENTIONS:
Behavioral: maternal education — Antenatal and/or postpartum Instruction on risks of neonatal jaundice, dangerous practices, technique to evaluate jaundice, early signs of ABE, when to seek care.
  Arms: maternal education

SUMMARY:
This study examines (a) whether introduction of public, health provider, and maternal education about risks of jaundice will decrease the occurrence of ABE compared with baseline prevalence (before-after design) or (b) whether antenatal or postpartum instruction to mothers will decrease the incidence of ABE compared with those who did not received instruction (concurrent opportunistic controls in phase 2).

DETAILED DESCRIPTION:
This 2 phase study first determines the prevalence of acute bilirubin encephalopathy (ABE) among newborns admitted for treatment of jaundice at 5 regional centers in Nigeria and identifies social/behavioral/medical factors associated with ABE. Information gained in phase 1 identified high risk sub-populations and guided selection of instructional materials for phase 2. Core data sheets submitted monthly by participating centers included clinical data, demographic information, number of antenatal clinic visits, birth place (hospital, clinic, home) and attendant, distance from care centers and reasons for delay, if any, in seeking care. Receipt of jaundice instruction by mothers is self-reported. Statistical analysis includes Chi square and logistic regression analysis of risk factors. Sample size: 1,000 subjects in each phase are required to demonstrate a 20% decrease in disease prevalence (baseline ABE incidence anticipated to be 15% of jaundiced babies) at 95% confidence level.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infant receiving treatment for neonatal jaundice

Exclusion Criteria:

* Non-viable premature infants
* Severe congenital defects.
* Postnatal age greater than 21 days

Ages: 30 Minutes to 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1765 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Acute bilirubin encephalopathy | at time of admission or discharge (1-21 days of life)
  Clinical signs of bilirubin toxicity described by unique neurological features in the presence of hyperbilirubinemia: reported as yes, no, or suspect (mild signs)

SECONDARY OUTCOMES:
Death from acute bilirubin encephalopathy or combined ABE/sepsis | 1-21 days of life
  Clinical signs of severe bilirubin toxicity with or without clinical signs of sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Oguche, MBBS, Study Director — Jos University Teaching Hospital; Abieyuwa Emokpae, MBBS, Study Director — Massey Street Pediatric Hospital, Lagos; Zubaida Farouk, MBBS, Study Director — Aminu Kano Teaching Hospital; Angela Okolo, MBBS, Study Director — Federal Medical Center Asaba; Isa Abdulkadir, MBBS, Study Director — Ahmadu Bello University Teaching Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Johnson L, Bhutani VK, Karp K, Sivieri EM, Shapiro SM. Clinical report from the pilot USA Kernicterus Registry (1992 to 2004). J Perinatol. 2009 Feb;29 Suppl 1:S25-45. doi: 10.1038/jp.2008.211. PMID 19177057
- [Result] Shapiro SM. Chronic bilirubin encephalopathy: diagnosis and outcome. Semin Fetal Neonatal Med. 2010 Jun;15(3):157-63. doi: 10.1016/j.siny.2009.12.004. Epub 2010 Jan 29. PMID 20116355